CLINICAL TRIAL: NCT02828111
Title: Double-Blind, Dose Escalating, Randomized, Vehicle-Controlled Proof of Concept Clinical Trial of Patidegib Gel 2%, 4%, and Vehicle Applied Once or Twice Daily to Decrease the GLI1 Biomarker in Sporadic Nodular Basal Cell Carcinomas
Brief Title: Clinical Trial of Patidegib Gel 2%, 4%, and Vehicle Applied Once or Twice Daily to Decrease the GLI1 Biomarker in Sporadic Nodular Basal Cell Carcinomas
Acronym: BCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PellePharm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pelle-926-202
Record Dates: First submitted 2016-07-01; First posted 2016-07-11 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Basal Cell Carcinomas
Keywords: Gorlin Syndrome; Basal Cell Nevus Syndrome BCNS; nevoid basal cell carcinoma syndrome; Basal cell carcinoma; Hedgehog inhibitor; Surgically Eligible Basal Cell Carcinomas; High Frequency Basal Cell Carcinomas
MeSH Terms: conditions — Carcinoma, Basal Cell; Basal Cell Nevus Syndrome | interventions — IPI-926; Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Patidegib gel 2% - Cohort 1 (Experimental): Patidegib gel 2%, applied topically, once daily for 12 weeks (Cohort 1)
  Interventions: Drug: Patidegib
- Patidegib gel 4% - Cohort 2 (Experimental): Patidegib gel 4%, applied topically, once daily for 12 weeks (Cohort 2)
  Interventions: Drug: Patidegib
- Vehicle gel - Cohort 1 (Placebo Comparator): Vehicle gel, applied topically, once daily for 12 weeks (Cohort 1)
  Interventions: Drug: Vehicle gel
- Patidegib gel 2% - Cohort 3 (Experimental): Patidegib gel 2%, applied topically, twice daily for 12 weeks (Cohort 3)
  Interventions: Drug: Patidegib
- Patidegib gel 4% - Cohort 4 (Experimental): Patidegib gel 4%, applied topically, twice daily for 12 weeks (Cohort 4)
  Interventions: Drug: Patidegib
- Vehicle gel - Cohort 2 (Placebo Comparator): Vehicle gel, applied topically, once daily for 12 weeks (Cohort 2)
  Interventions: Drug: Vehicle gel
- Vehicle gel - Cohort 3 (Placebo Comparator): Vehicle gel, applied topically, twice daily for 12 weeks (Cohort 3)
  Interventions: Drug: Vehicle gel
- Vehicle gel - Cohort 4 (Placebo Comparator): Vehicle gel, applied topically, twice daily for 12 weeks (Cohort 4)
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: Patidegib
  Other Names: Study drug
  Arms: Patidegib gel 2% - Cohort 1; Patidegib gel 2% - Cohort 3; Patidegib gel 4% - Cohort 2; Patidegib gel 4% - Cohort 4
Drug: Vehicle gel
  Other Names: Placebo
  Arms: Vehicle gel - Cohort 1; Vehicle gel - Cohort 2; Vehicle gel - Cohort 3; Vehicle gel - Cohort 4

SUMMARY:
This is a double-blind, dose escalating, randomized, vehicle-controlled study designed to compare the efficacy and safety of patidegib gel 2% and 4% applied once or twice daily in comparison with that of vehicle in patients with Basal Cell Carcinoma. One investigational center (metasite) in the United States will participate in this study. Approximately 36 subjects who meet the study entry criteria will be enrolled into one of four sequential cohorts. Within each cohort subjects will be randomized in a 2:1 ratio to receive active or vehicle gel.

DETAILED DESCRIPTION:
This is a double-blind, dose escalating, randomized, vehicle-controlled study designed to compare the efficacy and safety of patidegib gel 2% and 4% applied once or twice daily in comparison with that of vehicle. Approximately 36 subjects who meet the study entry criteria will be enrolled into one of four sequential cohorts. As soon as one cohort has been completely enrolled, the next cohort will be enrolled. Each subject will treat no more than two previously untreated biopsy confirmed treatment-targeted nodular BCCs. If the subject has additional non-treatment targeted BCCs they can be treated surgically prior to or during the trial. Within each cohort subjects will be randomized in a 2:1 ratio to receive active or vehicle gel. The sequential cohorts will be:

* Cohort 1: patidegib gel 2% or vehicle, once daily
* Cohort 2: patidegib gel 4% or vehicle, once daily
* Cohort 3: patidegib gel 2% or vehicle, twice daily
* Cohort 4: patidegib gel 4% or vehicle, twice daily

The study drug will be applied topically to the treatment-targeted BCCs and a rim of adjacent skin for 12 weeks. Information on reported and observed adverse events (AEs) will be obtained at each visit. An abbreviated physical examination (PE) will be performed at Baseline and Week 12. The treatment-targeted BCCs will be identified by the Investigator at the Baseline visit and will be circled in ink at Baseline, Weeks 6 and 12 and photographed, and measured at all study visits (Baseline, Weeks 2, 6, 8, 10, and 12). Blood samples for complete blood count and serum chemistry and urine for urinalysis will be collected from subjects at Screening, Week 6, and Week 12. Subjects who terminate study participation early will be asked to complete all Week 12 assessments, as appropriate, prior to commencement of any alternative therapy for BCCs (if possible). Subjects who discontinue from the study during the treatment period will not be replaced.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is from 18 to 85 years of age, inclusive.
2. The participant must provide electronic informed consent prior to any study procedures.
3. If the participant is a woman of childbearing potential, she is willing to use two effective methods of birth control during the duration of the trial and for one month after the last application of the gel. The two forms of birth control authorized are defined as the use of a barrier method of contraception (condom with spermicide) in association with one of the following methods of birth control: bilateral tubal ligation; combined oral contraceptives (estrogens and progesterone) or implanted or injectable contraceptives with a stable dose for at least 1 month prior to Baseline; hormonal intra-uterine device (IUD) inserted at least 1 month prior to Baseline. This proscription is based on the key role of the hedgehog (HH) pathway in embryogenesis, the known preclinical teratogenic effects of systemic cyclopamine, a naturally occurring inhibitor of smoothened (SMO), and the unknown level of systemic exposure following topical application of patidegib in humans.
4. If the participant is a male with a female sexual partner who is of childbearing potential, the couple is willing to use two effective methods of birth control during the duration of the trial and for one month after the last application of the gel. Authorized birth control methods are outlined in Inclusion Criterion #3. Any woman of childbearing potential applying the gel to themselves, or assisting a subject, must comply with the same birth control measures.
5. One or two previously untreated basal cell carcinomas (BCCs) with the clinical features of a nodular BCC confirmed by a biopsy done at or prior to screening confirming nodular BCC. These tumors must be suitable for surgical excision. The BCCs prior to biopsy must be no less than 5 millimeters (mm) or greater than 15 mm in greatest diameter on the face and no less than 9 mm or more than 20 mm in greatest diameter at sites other than the face. Tumors on the nose, periorbital skin, or on or below the knee are excluded.
6. The participant is willing to abstain from application of non-study topical prescription and over the counter medications within 5 centimeters (cm) of a treatment-targeted BCC for the duration of the study except as prescribed by the Investigator. Moisturizers and emollients are allowable. Subjects will be encouraged to use sunscreen with a sunscreen protection factor (SPF 15 or higher) at least once daily on all exposed skin sites.
7. Female participant must have negative serum pregnancy test at Screening.
8. The participant is willing to contact the study center after each primary skin care physician (PSCP) visit to provide the study center details of the visit and any treatment of skin tumors.
9. The participant is willing to forego alternative treatment of the treatment-targeted baseline BCC for the duration of the trial.

Exclusion Criteria:

1. Participants with basal cell nevus syndrome (BCNS, Gorlin syndrome, nevoid basal cell carcinoma syndrome; Online Mendelian Inheritance in Man [OMIM] #109400).
2. The participant has used topical products within 5 cm of a treatment- targeted BCC or systemic therapies that might interfere with the evaluation of the study medication during the study. Specifically, these include the use of:

   1. Topical glucocorticoids 30 days prior to screening
   2. Retinoids (such as etretinate, isotretinoin, tazarotene, tretinoin, adapalene) systemically or topically, or > 5% of an alphahydroxy acid (such as glycolic acid, lactic acid), photodynamic therapy (PDT), or 5-fluorouracil or imiquimod (except as topical treatment to discrete BCCs) systemically or topically to the skin during the six months prior to entry.
   3. Systemic chemotherapy within one year prior to screening. (Note: field therapy with topically applied treatments can be done as long as they are not applied within 5 cm of a treatment-targeted tumor).
   4. Known inhibitors of the HH signaling pathway (such as vismodegib, patidegib, sonidegib, and itraconazole) topically or systemically within 6 months of entry into the study.
3. The participant has a history of hypersensitivity to any of the ingredients in the study medication formulation.
4. The participant is unable or unwilling to make a good faith effort to be present for all follow-up visits and tests.
5. The participant is a woman who is currently nursing.
6. The participant has any systemic disease that in the Investigator's opinion would interfere with the subject's ability to participate.
7. The participant has a clinically significant history of liver disease, including viral hepatitis, current alcohol abuse, or cirrhosis, that in the investigator's opinion would interfere with the participant's ability to participate.
8. The participant has any condition or situation which in the Investigator's opinion may put the subject at significant risk, could confound the study results, or could interfere significantly with the participant's participation in the study. This includes history of other skin conditions or diseases, metabolic dysfunction, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that contraindicates use of this investigational drug or that might affect interpretation of the results of the study or render the participant at high risk from treatment complications.
9. The participant has a history of invasive cancer within the past five years excluding non-melanoma skin cancer, Stage I cervical cancer, ductal carcinoma in situ of breast, or chronic lymphocytic lymphoma (CLL) (Stage 0).
10. The participant is currently participating in an experimental drug study (within 4 weeks of Baseline visit) or plans to participate in an experimental drug study while enrolled in this study.
11. The participant is on a concomitant medication that is a strong CYP3A4 inhibitor. These include, but are not limited to: larithromycin, telithromycin, nefazodone, itraconazole, ketoconazole, atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, and tipranavir.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ervin Epstein, MD, Study Director — PellePharm, Inc.
Locations (1):
- 12121 Bluff Creek Drive Suite 100, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patidegib Gel 2% - Once Daily: Applied topically once daily for 12 weeks (Cohort 1)
- Patidegib Gel 4% - Once Daily: Applied topically once daily for 12 weeks (Cohort 2)
- Patidegib Gel 2% - Twice Daily: Applied topically twice daily for 12 weeks (Cohort 3)
- Patidegib Gel 4% - Twice Daily: Applied topically twice daily for 12 weeks (Cohort 4)
- Vehicle Gel: Applied topically once or twice daily for 12 weeks (Cohorts 1, 2, 3, and 4)
Period: Overall Study
Arm/Group | Patidegib Gel 2% - Once Daily | Patidegib Gel 4% - Once Daily | Patidegib Gel 2% - Twice Daily | Patidegib Gel 4% - Twice Daily | Vehicle Gel
Started | 6 | 6 | 6 | 6 | 12
Received at Least 1 Dose of Study Drug | 6 | 6 | 6 | 6 | 12
Completed | 6 | 6 | 4 | 5 | 11
Not Completed | 0 | 0 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Patidegib Gel 2% - Once Daily | Patidegib Gel 4% - Once Daily | Patidegib Gel 2% - Twice Daily | Patidegib Gel 4% - Twice Daily | Vehicle Gel | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (7.81) | 69.5 (12.32) | 64.7 (9.50) | 62.0 (7.85) | 63.9 (9.15) | 62.5 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 0 | 3 | 7 | 16
  Male | 2 | 4 | 6 | 3 | 5 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 12 | 36
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 12 | 36
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 86.43 (21.248) | 83.93 (14.901) | 99.50 (23.595) | 73.93 (10.874) | 83.76 (23.744) | 85.22 (20.69)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events (Including Both Serious and Non-Serious) Causally Related to Study Drug
Description: All serious adverse events (SAEs) and all other non-serious adverse events (AEs) regardless of causality are located in the Reported AE Module. The number of AEs (including both serious and non-serious) considered related to study drug by the Investigator are presented below. Treatment-emergent AEs are those with an onset after use of study drug.
Time Frame: Baseline through Week 12
Population: All enrolled participants who were randomized, received at least 1 confirmed dose of study drug, and had at least 1 post-baseline safety assessment.
Measure: Number; unit: number of events
Arm/Group | Patidegib Gel 2% - Once Daily | Patidegib Gel 4% - Once Daily | Patidegib Gel 2% - Twice Daily | Patidegib Gel 4% - Twice Daily | Vehicle Gel
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 12
number of events | 0 | 0 | 0 | 2 | 0

2. Primary Outcome: Molecular Efficacy: Percent Change From Baseline in the Hedgehog (HH) Signaling Pathway Target Gene Glioma-associated Oncogene Homolog 1 (GLI1) Messenger Ribonucleic Acid (mRNA) Levels at Week 12
Description: GLI1 change is a biomarker of the HH signaling pathway. A change in GLI1 mRNA levels reflect a change in the HH pathway. Surgically eligible basal cell carcinomas (SEBs) were defined as clinically diagnosed basal cell carcinoma (BCC) 5 to 20 millimeters (mm) in diameter on the face, excluding the nose and periorbital skin, and 9 to 20 mm at sites other than the face. A single baseline BCC designated as a treatment-targeted tumor at Baseline was biopsied first at Baseline and again following 12 weeks of treatment. This was used to assess percent change in GLI1 mRNA levels as follows: (Baseline - Week 12) / Baseline * 100, with positive numbers to represent increases and negative numbers to represent decreases. Any missing values were not imputed; all available data is summarized.
Time Frame: Baseline, Week 12
Population: Participants who received at least 1 dose of study drug who had evaluable GLI1 mRNA data at Baseline and Week 12.
Measure: Mean (Standard Deviation); unit: percent change in GLI1 mRNA levels
Arm/Group | Patidegib Gel 2% - Once Daily | Patidegib Gel 4% - Once Daily | Patidegib Gel 2% - Twice Daily | Patidegib Gel 4% - Twice Daily | Vehicle Gel
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
percent change in GLI1 mRNA levels | -56.300 (99.5901) | -3.243 (69.0247) | -42.510 (55.6352) | -28.847 (46.2318) | 23.306 (51.6076)
Statistical Analysis 1: Comparison: Patidegib Gel 2% - Once Daily vs Vehicle Gel; at Week 12; Test type: Other — Pairwise comparison; p = 0.132, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate
Statistical Analysis 2: Comparison: Patidegib Gel 4% - Once Daily vs Vehicle Gel; at Week 12; Test type: Other — Pairwise comparison; p = 0.658, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate
Statistical Analysis 3: Comparison: Patidegib Gel 2% - Twice Daily vs Vehicle Gel; at Week 12; Test type: Other — Pairwise comparison; p = 0.142, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate
Statistical Analysis 4: Comparison: Patidegib Gel 4% - Twice Daily vs Vehicle Gel; at Week 12; Test type: Other — Pairwise comparison; p = 0.207, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate
Statistical Analysis 5: Comparison: Patidegib Gel 2% - Once Daily vs Patidegib Gel 2% - Twice Daily vs Vehicle Gel; This is the analysis of combined patidegib gel 2% once daily and twice daily compared with vehicle gel at Week 12; Test type: Other — Pairwise comparison; p = 0.077, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate
Statistical Analysis 6: Comparison: Patidegib Gel 4% - Once Daily vs Patidegib Gel 4% - Twice Daily vs Vehicle Gel; This is the analysis of combined patidegib gel 4% once daily and twice daily compared with vehicle gel at Week 12; Test type: Other — Pairwise comparison; p = 0.331, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate
Statistical Analysis 7: Comparison: Patidegib Gel 2% - Once Daily vs Patidegib Gel 4% - Once Daily vs Patidegib Gel 2% - Twice Daily vs Patidegib Gel 4% - Twice Daily vs Vehicle Gel; This is the analysis of all four patidegib gel treatment groups combined compared with vehicle gel at Week 12; Test type: Other — Pairwise comparison; p = 0.117, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate

3. Secondary Outcome: Clinical Efficacy: Percent Change From Baseline in Tumor Size of Treatment-targeted SEBs at Week 12
Description: SEBs were defined as clinically diagnosed BCC 5 to 20 mm in diameter on the face, excluding the nose and periorbital skin, and 9 to 20 mm at sites other than the face. The percent change in greatest diameters of treatment-targeted surgically eligible basal cell carcinomas (SEBs) from Baseline to Week 12 was calculated as follows: (sum [Baseline] - sum [Week 12] / sum [Baseline] * 100), where sum = the greatest diameters of treatment-targeted SEBs and positive numbers to represent increases and negative numbers to represent decreases. Missing values were imputed using Last-Observation Carried Forward (LOCF).
Time Frame: Baseline, Week 12
Population: Participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percent change in tumor size
Arm/Group | Patidegib Gel 2% - Cohort 1 | Vehicle Gel - Cohort 1 | Patidegib Gel 4% - Cohort 2 | Vehicle Gel - Cohort 2 | Patidegib Gel 2% - Cohort 3 | Vehicle Gel - Cohort 3 | Patidegib Gel 4% - Cohort 4 | Vehicle Gel - Cohort 4
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 6 | 3 | 6 | 3
percent change in tumor size | 56.15 (48.138) | 5.08 (33.541) | 8.73 (46.600) | 51.11 (60.584) | 17.01 (36.870) | 51.11 (42.861) | 18.41 (60.592) | 33.33 (57.735)

4. Secondary Outcome: Clinical Efficacy: Percentage of SEBs Showing Complete or Partial Response at Week 12 as Determined by Blinded Photographic Review
Description: SEBs were defined as clinically diagnosed BCC 5 to 20 mm in diameter on the face, excluding the nose and periorbital skin, and 9 to 20 mm at sites other than the face. The percentage of tumors showing a complete or partial response at Week 12 was calculated as follows: (Number of baseline treatment-targeted SEBs showing complete or partial response at Week 12) / (Number of Baseline treatment-targeted SEBs) * 100. Missing values were not imputed.Complete Response is determined when there is no longer any visible evidence of a lesion consistent with BCC at the site, and Partial Response is determined when although a BCC still remains at this site, it has demonstrated a visible decrease in size compared with baseline.
Time Frame: Baseline, Week 12
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of SEBs
Arm/Group | Patidegib Gel 2% - Cohort 1 | Vehicle Gel - Cohort 1 | Patidegib Gel 4% - Cohort 2 | Vehicle Gel - Cohort 2 | Patidegib Gel 2% - Cohort 3 | Vehicle Gel - Cohort 3 | Patidegib Gel 4% - Cohort 4 | Vehicle Gel - Cohort 4
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 6 | 3 | 6 | 3
percentage of SEBs | 71.4 | 0 | 50.0 | 100 | 25.0 | 100 | 66.7 | 50.0

5. Other Pre Specified Outcome: Percentage of Treatment-targeted SEBs Achieving Clear or Almost Clear on the Investigator Static Global Tumor Assessment (ISGTA) Scale
Description: The ISGTA is a scale with scores ranging from 0 (clear), 1 (almost clear), 2 (minimal residual tumor), to 3 (clearly visible tumor). The Investigator assessed each Baseline treatment-targeted SEB at Weeks 2, 6, 8, 10, and 12. SEBs were defined as clinically diagnosed BCC 5 to 20 mm in diameter on the face, excluding the nose and periorbital skin, and 9 to 20 mm at sites other than the face. The percentage of Baseline treatment-targeted SEBs evaluated as being clear or almost clear at Week x (Week x = 2, 6, 8, 10, or 12) based on the ISGTA scale was calculated as follows: (Number of baseline treatment-targeted SEBs with ISGTA score of 0 or 1 at Week x) / (Number of Baseline treatment-targeted SEBs) * 100. Missing data were imputed using LOCF. The percentage of responders achieving clear (0) or almost clear (1) on the ISGTA scale are presented by Week.
Time Frame: Baseline and Weeks 2, 6, 8, 10, and 12
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of SEBs
Arm/Group | Patidegib Gel 2% - Cohort 1 | Vehicle Gel - Cohort 1 | Patidegib Gel 4% - Cohort 2 | Vehicle Gel - Cohort 2 | Patidegib Gel 2% - Cohort 3 | Vehicle Gel - Cohort 3 | Patidegib Gel 4% - Cohort 4 | Vehicle Gel - Cohort 4
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 6 | 3 | 6 | 3
percentage of SEBs
  Week 2 | 14.3 | 0 | 0 | 33.3 | 28.6 | 0 | 0 | 0
  Week 6 | 14.3 | 0 | 0 | 33.3 | 14.3 | 0 | 16.7 | 0
  Week 8 | 14.3 | 0 | 0 | 33.3 | 14.3 | 0 | 16.7 | 0
  Week 10 | 42.9 | 0 | 0 | 66.7 | 28.6 | 33.3 | 16.7 | 33.3
  Week 12 | 57.1 | 0 | 16.7 | 33.3 | 14.3 | 33.3 | 16.7 | 33.3

6. Other Pre Specified Outcome: Percent Change in Treatment-targeted SEBs Tumor Size From Baseline as Determined by Blinded Photographic Review
Description: SEBs were defined as clinically diagnosed BCC 5 to 20 mm in diameter on the face, excluding the nose and periorbital skin, and 9 to 20 mm at sites other than the face. The percent change in greatest diameters of Baseline treatment-targeted SEBs from Baseline to Week 12 was calculated as follows: (sum [Baseline] - sum [Week 12] / sum [Baseline]) * 100), where sum = the greatest diameters of treatment-targeted SEBs.
Time Frame: Baseline, Week 12
Population: Participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage change from Baseline
Arm/Group | Patidegib Gel 2% - Cohort 1 | Vehicle Gel - Cohort 1 | Patidegib Gel 4% - Cohort 2 | Vehicle Gel - Cohort 2 | Patidegib Gel 2% - Cohort 3 | Vehicle Gel - Cohort 3 | Patidegib Gel 4% - Cohort 4 | Vehicle Gel - Cohort 4
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 6 | 3 | 6 | 3
percentage change from Baseline | -43.464 (55.7676) | 24.995 (32.3747) | -3.686 (37.8650) | 46.095 (97.4129) | -13.462 (60.7358) | -69.518 (52.7961) | -25.836 (45.5819) | -26.481 (59.9186)
Statistical Analysis 1: Comparison: Patidegib Gel 2% - Cohort 1 vs Vehicle Gel - Cohort 1; at Week 12; Test type: Other — Pairwise comparison; p = 0.038, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate
Statistical Analysis 2: Comparison: Patidegib Gel 4% - Cohort 2 vs Vehicle Gel - Cohort 2; at Week 12; Test type: Other — Pairwise comparison; p = 0.099, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate
Statistical Analysis 3: Comparison: Patidegib Gel 2% - Cohort 3 vs Vehicle Gel - Cohort 3; at Week 12; Test type: Other — Pairwise comparison; p = 0.198, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate
Statistical Analysis 4: Comparison: Patidegib Gel 4% - Cohort 4 vs Vehicle Gel - Cohort 4; at Week 12; Test type: Other — Pairwise comparison; p = 0.757, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate

7. Post Hoc Outcome: Percentage of Treatment-targeted SEBs Achieving Clear on the ISGTA Scale and BCC Not Present at Week 12
Description: The ISGTA is a scale with scores ranging from 0 (clear), 1 (almost clear), 2 (minimal residual tumor), to 3 (clearly visible tumor). The Investigator assessed each Baseline treatment-targeted SEB at Week 12. SEBs were defined as clinically diagnosed BCC 5 to 20 mm in diameter on the face, excluding the nose and periorbital skin, and 9 to 20 mm at sites other than the face. The percentage of Baseline treatment-targeted SEBs evaluated as being clear at Week 12 based on the ISGTA scale and BCC not present was calculated as follows: (Number of baseline treatment-targeted SEBs with ISGTA score of 0 and BCC not present at Week 12) / (Number of Baseline treatment-targeted SEBs) * 100.
Time Frame: Week 12
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of SEBs
Groups:
- Vehicle Gel - All Cohorts: Vehicle gel, applied topically once or twice daily for 12 weeks (Cohorts 1, 2, 3, and 4)
Arm/Group | Patidegib Gel 2% - Cohort 1 | Vehicle Gel - Cohort 1 | Patidegib Gel 4% - Cohort 2 | Vehicle Gel - Cohort 2 | Patidegib Gel 2% - Cohort 3 | Vehicle Gel - Cohort 3 | Patidegib Gel 4% - Cohort 4 | Vehicle Gel - Cohort 4 | Vehicle Gel - All Cohorts
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 6 | 3 | 6 | 3 | 12
percentage of SEBs | 42.9 | 0 | 0 | 0 | 20.0 | 0 | 16.7 | 0 | 0
Statistical Analysis 1: Comparison: Patidegib Gel 2% - Cohort 1 vs Vehicle Gel - All Cohorts; at Week 12; Test type: Other — Pairwise comparison; p = 0.043, Fisher Exact
Statistical Analysis 2: Comparison: Patidegib Gel 2% - Cohort 3 vs Vehicle Gel - All Cohorts; at Week 12; Test type: Other — Pairwise comparison; p = 0.312, Fisher Exact
Statistical Analysis 3: Comparison: Patidegib Gel 4% - Cohort 4 vs Vehicle Gel - All Cohorts; at Week 12; Test type: Other — Pairwise comparison; p = 0.353, Fisher Exact
Statistical Analysis 4: Comparison: Patidegib Gel 2% - Cohort 1 vs Patidegib Gel 2% - Cohort 3 vs Vehicle Gel - All Cohorts; This is the analysis of combined patidegib gel 2% once daily and twice daily compared with vehicle gel at Week 12; Test type: Other — Pairwise comparison; p = 0.093, Fisher Exact
Statistical Analysis 5: Comparison: Patidegib Gel 4% - Cohort 2 vs Patidegib Gel 4% - Cohort 4 vs Vehicle Gel - All Cohorts; This is the analysis of combined patidegib gel 4% once daily and twice daily compared with vehicle gel at Week 12; Test type: Other — Pairwise comparison; p = 1.000, Fisher Exact
Statistical Analysis 6: Comparison: Patidegib Gel 2% - Cohort 1 vs Patidegib Gel 4% - Cohort 2 vs Patidegib Gel 2% - Cohort 3 vs Patidegib Gel 4% - Cohort 4 vs Vehicle Gel - All Cohorts; This is the analysis of all four patidegib gel treatment groups combined compared with combined vehicle gel at Week 12; Test type: Other — Pairwise comparison; p = 0.157, Fisher Exact

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: All enrolled participants who were randomized, received at least 1 confirmed dose of study drug, and had at least 1 post-baseline safety assessment.
Arm/Group | Patidegib Gel 2% - Once Daily | Patidegib Gel 4% - Once Daily | Patidegib Gel 2% - Twice Daily | Patidegib Gel 4% - Twice Daily | Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/6 | 1/12
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 1/5 | 3/6 | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patidegib Gel 2% - Once Daily (N=6) | Patidegib Gel 4% - Once Daily (N=6) | Patidegib Gel 2% - Twice Daily (N=5) | Patidegib Gel 4% - Twice Daily (N=6) | Vehicle Gel (N=12)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patidegib Gel 2% - Once Daily (N=6) | Patidegib Gel 4% - Once Daily (N=6) | Patidegib Gel 2% - Twice Daily (N=5) | Patidegib Gel 4% - Twice Daily (N=6) | Vehicle Gel (N=12)
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Application site oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuromuscular pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT02828111/SAP_000.pdf
  • Study Protocol (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT02828111/Prot_001.pdf